CLINICAL TRIAL: NCT00271934
Title: Immune Ablation and Hematopoietic Stem Cell Support in Patients With Poor Prognostic Indicators and Systemic Lupus Erythematosus:A Phase II Study
Brief Title: Immune Ablation and Hematopoietic Stem Cell Support in Patients With Systemic Lupus Erythematosus: A Phase II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU95LU1
Record Dates: First submitted 2006-01-02; First posted 2006-01-04 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Immune ablation and hematopoietic stem cell support. — Autologous hematopoietic stem cell transplant

SUMMARY:
In patients with systemic lupus erythematosus, immunosuppressive therapy to the point of complete immune ablation and hematopoietic stem cell recovery.

DETAILED DESCRIPTION:
Systemic lupus erythematosus is a multisystem, inflammatory disorder characterized by the production of antibodies that react with many different self-antigens. Defects in immune regulation underlie the breakdown in self-tolerance.(1) The clinical course of lupus is variable. Aggressive intervention is reserved for disease with characteristic high risk features including diffuse, proliferative glomerulonephritis, pulmonary hemorrhage, cerebritis and other life-threatening manifestations of vasculitis. In patients with SLE and high risk features, we propose extension of current immunosuppressive therapy to the point of complete immune ablation and hematopoietic stem cell recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Less than age of 60 year at the time of pretransplant evaluation.
2. An established clinical diagnosis of systemic lupus erythematosus with one of the following features:

   1. Lupus nephritis-WHO class III or IV (or V when coexistent III or IV) lupus nephritis, failing NIH short course cyclophosphamide therapy (10mg/kg q month for 6 months). Failure will be defined as failure of creatinine to return to normal or pre-exacerbation level.
   2. Vasculitis/Immune complex deposition- causing end organ signs or symptoms e.g. cerebritis, transverse myelitis, pulmonary hemorrhage, cardiac failure, renal failure.
   3. Cytopenias that are immune-mediated and not controlled by conservative measures including danzole, prednisone, and alkylating agents (cyclophosphamide or vincristine); and any one of the following: transfusion dependant anemia with untransfused hemoglobin less than 8 grams/dl, or platelets less than 40,000/ul without transfusions,or granulocytes less than 1000/ul.
   4. Catastrophic Anti-phospholipid Syndrome

4. Ability and willingness to provide informed consent.

Exclusion Criteria:

1. Human immunodeficiency virus (HIV)positive status.
2. History of unstable angina.
3. Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemoradiotherapy.
4. Prior history of malignancy except for localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as head and neck cancer, or stage I breast cancer will be considered on an individual basis.
5. Positive serum pregnancy test, inability or unwillingness to pursue effective means of birth control or failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
6. Psychiatric illness or mental deficiency not due to active lupus cerebritis making compliance with treatment or informed consent impossible.
7. FEV1/FVC<50% of predicted, DLCO <50%of predicted.
8. Resting left ventricular ejection fraction(LVEF)<35% or lupus induced myocarditis.
9. Known hypersensitivity to Escherichia coli.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2002-09; Primary Completion 2007-11 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
SLEDAI | 5 years after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Result] Burt RK, Traynor A, Statkute L, Barr WG, Rosa R, Schroeder J, Verda L, Krosnjar N, Quigley K, Yaung K, Villa Bs M, Takahashi M, Jovanovic B, Oyama Y. Nonmyeloablative hematopoietic stem cell transplantation for systemic lupus erythematosus. JAMA. 2006 Feb 1;295(5):527-35. doi: 10.1001/jama.295.5.527. PMID 16449618